CLINICAL TRIAL: NCT03274167
Title: Efficacy of Gabapentin in Alcohol Dependency Treatment: a Double-blinded Randomized Placebo-controlled Trial
Brief Title: Efficacy of Gabapentin in Alcohol Dependency Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Princess Mother National Institute on Drug Abuse and Treatment (Unknown)
Responsible Party: Principal Investigator, Rasmon Kalayasiri, Associate Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: PMNIDAT#xx/2012
Record Dates: First submitted 2017-08-29; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Alcohol Drinking; Heavy Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Gabapentin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Experimental): 300 mg per day once daily before bedtime
  Interventions: Drug: Gabapentin 300mg
- Control (Placebo Comparator): Capsule identical to the experimental arm, one tablet once daily before bedtime
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Gabapentin 300mg
  Arms: Gabapentin
Drug: Placebo oral capsule
  Arms: Control

SUMMARY:
The study aims to study the effect of gabapentin on the number of alcohol drinking days and heavy drinking days in the Thai clinical alcohol-dependent population by using the double-blinded randomized controlled approach. One-hundred and twelve individuals with alcohol dependence were randomly assigned equally into two groups including treatment with gabapentin and placebo. Thirty-four patients (30.3%) completed the study protocol, i.e. treatment with gabapentin at least 300 mg per day or placebo orally once a day for twelve weeks. Pattern of alcohol drinking were obtained from the timelime followback. Drinking behaviors were compared between the two groups by poisson repeated measures model.

ELIGIBILITY:
Inclusion Criteria:

* current diagnosis of alcohol dependence

Exclusion Criteria:

* having major psychiatric disorders including schizophrenia, schizoaffective disorder, bipolar disorder, major depressive disorder, or suicide risk based on a clinical interview by attending psychiatrist
* receiving other medications not in the protocol of the study for any reasons or having history of using other substances including methamphetamine, heroin, cannabis, inhalants, mitragyna speciosa (or kratom in Thai), except tobacco based on self-report
* having a medical disease, e.g. essential hypertension, diabetes, renal (e.g., normal renal test) or liver disease (e.g., liver function test was not higher than two times of normal range and gamma-glutamyl transferase (GGT) is less than 800 U/L), epilepsy, stroke
* having history of alcohol withdrawal seizure or delirium based on clinical interview by attending psychiatrist
* having moderate to severe alcohol withdrawal symptoms based on score >13 of the Clinical Interview for Withdrawal Alcohol Arlington (CIWA - Ar) at the time of recruitment
* having cognitive impairment based on score < 24 from the Mini Mental State Exam (MMSE)
* having history of allergy to gabapentin
* pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Frequency of heavy drinking | weekly for 12 weeks
  Days per week of alcohol heavy drinking as measured by timelime followback (TLFB) (Sobell et al., 2001) - adapted Thai version. TLFB is the self-report form for a respondent to note days of heavy alcohol drinking, daily amount, and any symptoms related to alcohol drinking including days per week of alcohol drinking. The TLFB was given to the subjects after explaining how to record daily drinking behaviors and symptoms at home.

SECONDARY OUTCOMES:
Frequency of drinking | weekly for 12 weeks
  Days per week of alcohol drinking as measured by timelime followback (TLFB) (Sobell et al., 2001) - adapted Thai version. TLFB is the self-report form for a respondent to note days of heavy alcohol drinking, daily amount, and any symptoms related to alcohol drinking including days per week of alcohol drinking. The TLFB was given to the subjects after explaining how to record daily drinking behaviors and symptoms at home.

CONTACTS AND LOCATIONS:
Overall Officials: Sumnao Nilaban, Principal Investigator — Princess Mother National Institute on Drug Abuse and Treatment
Locations (1):
- Princess Mother National Institute on Drug Abuse and Treatment, Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Undecided